CLINICAL TRIAL: NCT06144944
Title: Neoadjuvant Pyrotinib Combined With Chemotherapy Versus Chemotherapy in HR-positive/HER2-low (IHC 2+/FISH-negative) High-risk Early Breast Cancer: an Open-lable, Multi-center, Randomized Phase III Trial
Brief Title: Neoadjuvant Pyrotinib in HR-positive and HER2-low High-risk Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chang Gong, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PILHLE-002
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Invasive; Hormone-receptor-positive Breast Cancer; HER2 Low Breast Carcinoma; Early-stage Breast Cancer
Keywords: pyrotintb; HER2-low EBC; neoadjuvant; HR-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Epirubicin; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant pyrotinib combined with chemotherapy (Experimental)
  Interventions: Drug: Pyrotinib, epirubicin or doxorubicin, cyclophosphamide, paclitaxel
- Neoadjuvant chemotherapy (Placebo Comparator)
  Interventions: Drug: Epirubicin or doxorubicin, cyclophosphamide, paclitaxel

INTERVENTIONS:
Drug: Pyrotinib, epirubicin or doxorubicin, cyclophosphamide, paclitaxel — Pyrotinib 320 mg orally once daily, and epirubicin 90 mg/m² or doxorubicin 60 mg/m² plus cyclophosphamide 600 mg/m² intravenously on day 1 for four 3-week cycles followed by paclitaxel 175 mg/m² intravenously on day 1 or four 3-week cycles.
  Arms: Neoadjuvant pyrotinib combined with chemotherapy
Drug: Epirubicin or doxorubicin, cyclophosphamide, paclitaxel — Epirubicin 90 mg/m² or doxorubicin 60 mg/m² plus cyclophosphamide 600 mg/m² intravenously on day 1 for four 3-week cycles followed by paclitaxel 175 mg/m² intravenously on day 1 or four 3-week cycles.
  Arms: Neoadjuvant chemotherapy

SUMMARY:
This is a multi-center, open-lable, prospective, randomized phase III clinical trial to further validate the efficacy and safety of neoadjuvant pyrotinib combined with chemotherapy in HR-positive/HER2-low (IHC 2+/FISH-negative) high-risk early breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Must participate voluntarily, sign the informed consent form, and have good compliance
* Aged ≥ 18 and ≤ 70 years old with ECOG PS score of 0-1
* Histopathological newly diagnosed, unilateral, primary invasive breast cancer
* Histopathological hormone receptor-positve ( estrogen receptor and/or progesterone receptor ≥ 10% stained cells) and HER2-low (immunochemistry 2+ with fluorescent in situ hybridization negative)
* TNM stage-IIb/III, or TNM stage-IIa with high risk (N+, G3, or MammaPrint High-risk)
* At least one evaluable target breast lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Left ventricular ejection fraction ≥ 55%, Fridericia-corrected QT interval < 450 ms in males and < 470 ms in females
* White blood cell count: ≥ 3.0 × 10^9/L, absolute neutrophil count: ≥ 1.5 × 10^9/L, platelet count: ≥ 100 × 10^9/L, hemoglobin: ≥ 90 g/L
* Aspartate aminotransferase and alanine aminotransferase: ≤ 2.5 × ULN, alkaline phosphatase: ≤ 2.5 × ULN, blood total bilirubin: ≤ 1.5 × ULN, serum creatinine: ≤ 1.5 × ULN
* Non-menopausal or non-surgically sterilized female patients identified as non-pregnant and non-lactating and consented to contraception both during the trial and within 6 months after the last administration of the test drug

Exclusion Criteria:

* Metastatic BC, bilateral BC, occult BC, inflammatory BC, or with other malignant tumors
* Known history of hypersensitivity to the study drugs
* Patients who need receive other anti-tumor treatments (except for OFS) during neoadjuvant therapy as judged by the investigators
* With severe cardiac disease or discomfort that is not expected to tolerate treatment, including but not limited to: a) arrhythmia that requires medication or is clinically significant, or high-grade atrioventricular block, b) unstable angina, myocardial infarction, heart failure or clinically significant heart valve disease, c) poorly controlled hypertension or any heart disease unsuitable for participation in this trial as determined by the investigators
* Patients who participated in a clinical trial of another drug within 4 weeks prior to randomization or underwent BC-free surgery within 4 weeks or had not fully recovered after BC-free surgery
* Other malignancy in the past 5 years, other than cured cervical carcinoma in situ, basal or squamous cell carcinoma of skin
* Patients who had basic gastrointestinal diseases (especially long-term history of diarrhea or/and constipation), inability to swallow, intestinal obstruction or other factors will affect drugs administration and absorption
* Presence of accompanying diseases that may pose serious risks to the safety of the patient or may affect the patient's ability to complete the study (including but not limited to severe diabetes mellitus, active infection, thyroid disorders, etc.) as judged by the investigator
* With a history of immunodeficiency, including acquired or congenital immunodeficiencies, or a history of organ transplantation
* Past history of confirmed neurological or mental disorders, including epilepsy or dementia
* Other conditions of the subject determined by the investigator to be unsuitable for the study

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Residual Cancer Burden 0/1 rate as assessed by independent central review | Within 4 weeks after surgery
  The proportion of patients with RCB 0/I after neoadjuvant therapy according to the online Residual Cancer Burden Calculator provided by the MD Anderson Cancer Center as assessed by independent central review

SECONDARY OUTCOMES:
Residual Cancer Burden 0/1 rate as assessed by local pathology review | Within 4 weeks after surgery
  The proportion of patients with RCB 0/I after neoadjuvant therapy according to the online Residual Cancer Burden Calculator provided by the MD Anderson Cancer Center as assessed by local pathology review
Pathological complete response rate | Within 4 weeks after surgery
  The proportion of patients with no residual invasive tumor cells in the breast and axillary nodes, regardless of ductal carcinoma in situ
Objective response rate | Within 2 weeks of breast MR examination
  The percentage of patients who achieved a complete or partial response in breast according to the RECIST, version 1.1, based on MRI, at the end of cycle 2 neoadjuvant therapy and at the end of cycle 8 neoadjuvant therapy
Breast conservation surgery rate | Within 4 weeks after surgery
  The proportion of patients who had successful breast conservation surgery after neoadjuvant therapy
Health-related Quality of Life 1 | Within 7 days before the first treatment and the end of each cycle (each cycle is 21 days)
  The score of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (version 3)
Health-related Quality of Life 2 | Within 7 days before the first treatment and the end of each cycle (each cycle is 21 days)
  The score of Breast Cancer-Specific Module (QLQ-BR23)
5-year event-free survival | During the 5 years after random assignment
  the time from random assignment until any relapse, unequivocal tumor progression, or any-cause death
5-year overall survival | During the 5 years after random assignment
  the time from random assignment until any-cause death
Safety (AEs+SAEs) | from signing the informed consent form until 2 years after completion of neoadjuvant treatment
  General safety will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0). Ovarian toxicity will be evaluated by menstrual status and FSH and E2
Biomarkers (Immune cell subpopulations quantities) | Within 4 weeks after surgery
  The association between immune cell subpopulations quantities and RCB

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gong, Prof, Principal Investigator — Breast Tumor Center, Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in future research article after de-identification and the study protocol will be shared beginning 3 months and ending 5 years following publication. Proposals should be directed to gchang@mail.sysu.edu.cn and data will be shared by email
Supporting Information: Study Protocol
Time Frame: beginning 3 months and ending 5 years following publication of future research article
Access Criteria: Researchers who provide a methodologically sound proposal, that need to be approved by an approved accredited ethics committee